CLINICAL TRIAL: NCT06247774
Title: Reducing Heart Failure Risk in Late-Life With Physical Activity: Impact on Cardiac Structure and Function and Proteomic Signatures
Brief Title: Reducing Heart Failure Risk in Late-Life With Physical Activity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Sheila M. Hegde, MD, Principal Investigator, Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023p002781
Record Dates: First submitted 2024-01-23; First posted 2024-02-08 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Hypertension; Exercise Training; Cardiac Rehabilitation; Proteomics
MeSH Terms: conditions — Hypertension | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac Rehabilitation (Experimental): Participants will participate in a 12-week cardiac rehabilitation program
  Interventions: Behavioral: Cardiac Rehabilitation
- Attention Control (Placebo Comparator): Participants will not participate in a cardiac rehabilitation program and will receive phone calls in place of cardiac rehabilitation visits.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Cardiac Rehabilitation — Participation in a 12-week cardiac rehabilitation program
  Arms: Cardiac Rehabilitation
Behavioral: Attention Control — Participants will receive regular phone calls in place of cardiac rehabilitation visits
  Arms: Attention Control

SUMMARY:
The goal of this clinical trial is to learn about the molecular pathways associated with the benefit of a regular exercise program in patients with high blood pressure and who don't already participate in regular exercise.

The main question it aims to answer is to identify protein signatures associated with the benefits of a cardiac rehabilitation exercise program.

The trial will enroll 42 participants, who will be randomized to a 12 week cardiac rehabilitation exercise program versus control arm and asked to participate in the following at the beginning and end of study:

* Cardiopulmonary exercise test (CPET)
* Echocardiogram
* Physical function test
* 6-minute walk test
* Hand grip strength
* Quality of life questionnaire
* Blood draws

Researchers will compare results between those who do and don't participate in the exercise program.

DETAILED DESCRIPTION:
Lifestyle modification with physical activity (PA) appears to be protective of several age-related cardiovascular (CV) outcomes, including heart failure (HF), in a dose-dependent manner. While many studies with exercise training have demonstrated improvement in quality of life and cardiorespiratory fitness, findings have not been consistent with regards to the potential for exercise to preserve or even improve cardiac function in adults with HF. There remains incomplete understanding of the molecular pathways by which PA mitigates HF risk. Furthermore, exercise studies often exclude older adults, who are disproportionately affected by HF, though our preliminary data suggest the protective effects of PA extend to late-life. Older adults are at particularly heightened risk for HF with preserved ejection fraction (HFpEF), which is characterized by impaired left ventricular (LV) diastolic function and impaired systolic deformation despite preserved LV ejection fraction (LVEF). Unlike with HF with reduced ejection fraction (HFrEF), effective pharmacologic therapies or interventions to improve cardiac function among individuals with preserved LVEF are limited. Thus, there is a critical need to define the cardiovascular mechanisms by which PA impacts HF risk in older adults that may enable the identification of novel therapeutic targets to prevent HF and HFpEF in particular.

As proteins orchestrate and carry out cellular functions in health and in diseases, one method of characterizing changes in CV function is to investigate cell signaling by studying the circulating proteome. Proteomic approaches have previously been used to identify pathways relevant to myocardial infarction and have also been used to investigate molecular pathways characterizing PA and CV disease. A recent study demonstrated upregulation of inflammation-related proteins in HFpEF patients (n=228) compared to controls, and their association with worse indices of cardiac function. Specific proteomic patterns have also been associated with aerobic exercise, with 2 proteomic modules that were specifically preserved with aging in habitual exercisers. Data from Swedish cohorts has also shown an association of leisure-time PA with 28 CV-specific proteins involved in atherosclerotic processes. Serial multi-omic measures (including proteomics) have been used to demonstrate marked intra-individual changes in circulating proteins with acute exercise. More recently, high-throughput proteomic profiling has been successfully employed in younger adults to identify baseline protein levels associated with change in cardiorespiratory fitness following an exercise intervention. However, to-date, limited data exist regarding intervention-related changes in the proteome in older adults at risk for HF and the extent to which these changes correlate with changes in cardiorespiratory fitness.

Supervised exercise-training with cardiac rehabilitation (CR) has been well established as an effective method to improve maximal oxygen consumption (VO2 max), a measure of cardiorespiratory fitness. Improvement in VO2 max has also been demonstrated with exercise training in sedentary older adults over 65 years of age.

The objective of this proposal is to identify protein signatures characterizing the known benefits of a structured CR program on VO2 max. Our working hypotheses is that proteomic approaches will identify novel biomarkers that uniquely characterize molecular pathways associated with exercise training and CR-related changes in proteins will correlate with changes in VO2 max. Successful completion of this aim will identify possible novel protein signatures underlying the protective biological pathways mediated by a structured CR program that may be used as preliminary data for future grant proposals.

Aim: Identify molecular pathways underlying the beneficial effect of a structured PA intervention on functional capacity with the use of plasma proteomics in older sedentary adults at high risk of HF. (BWH-based cohort). Hypotheses: (1) Randomization to participation in a cardiac rehabilitation (CR) program will result in improvement in circulating levels of 4 plasma proteins associated with change in VO2max, a measure of cardiorespiratory fitness, and with genetic evidence supporting a causal effect on HF and cardiac structure (ATF6, STC1, JAG1, PTK7). The investigators will randomize 42 sedentary adults at high risk of HF (stage B HF) to participation in a CR program and perform proteomic analysis, cardiopulmonary exercise testing, and echocardiography at baseline and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension (controlled on stable medication regimen)
* Structural heart abnormality (LVH or LA enlargement)
* LVEF > 50%
* Sedentary
* BMI <30

Exclusion Criteria:

* Diabetes
* Unable to exercise
* Supplemental oxygen use
* Pulmonary hypertension
* Sleep apnea
* Regular exercise training
* Devices that limit ability to achieve target heart rate
* Moderate to severe valve disease
* Recent (within 3 months) major CV event or planned procedures (within 6 months)
* Terminal illness, life expectancy <6 months
* Inability or unwillingness to comply with study requirements
* No access to smart phone/tablet

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Impact of Cardiac Rehabilitation training on single protein changes | 12 weeks
  Change in protein levels assessed by blood draws and measured by Somascan assay. ANCOVA analysis adjusting for baseline protein levels with intention to treat group assignment

SECONDARY OUTCOMES:
Correlation of change in proteins with change in VO2 max | 12 weeks
  Correlation of single protein changes associated with change in VO2 max
Correlation of change in proteins with change in LV global longitudinal strain | 12 weeks
  Correlation of single protein changes associated with change in LV global longitudinal strain
Correlation of change in proteins with change in LV diastolic function | 12 weeks
  Correlation of single protein changes associated with change in LV diastolic function
Correlation of change in proteins with change in VE/VCO2 | 12 weeks
  Correlation of single protein changes associated with change in VE/VCO2
Correlation of change in proteins with change in Short Physical Performance Battery (SPPB) | 12 weeks
  Correlation of single protein changes associated with change in Short Physical Performance Battery (SPPB)
Correlation of change in proteins with change in 6-minute walk test | 12 weeks
  Correlation of single protein changes associated with change in 6-minute walk test
Correlation of change in proteins with change in grip strength | 12 weeks
  Correlation of single protein changes associated with change in grip strength
Correlation of change in proteins with change in EQ-5D (QOL) | 12 weeks
  Correlation of single protein changes associated with change in EQ-5D (QOL)
Correlation of change in proteins with change in step counts | 12 weeks
  Correlation of single protein changes associated with change in step counts
Correlation of baseline proteins with change in VO2 max | 12 weeks
  Correlation of baseline proteins with change in VO2 max
Correlation of baseline proteins with change in LV global longitudinal strain | 12 weeks
  Correlation of baseline proteins with change in LV global longitudinal strain
Correlation of baseline proteins with change in LV diastolic function | 12 weeks
  Correlation of baseline proteins with change in LV diastolic function
Correlation of baseline proteins with change in VE/VCO2 | 12 weeks
  Correlation of baseline proteins with change in VE/VCO2
Correlation of baseline proteins with change in SPPB | 12 weeks
  Correlation of baseline proteins with change in SPPB
Correlation of baseline proteins with change in 6-minute walk test | 12 weeks
  Correlation of baseline proteins with change in 6-minute walk test
Correlation of baseline proteins with change in grip strength | 12 weeks
  Correlation of baseline proteins with change in grip strength
Correlation of baseline proteins with change in EQ-5D (QOL) | 12 weeks
  Correlation of baseline proteins with change in EQ-5D (QOL)
Correlation of baseline proteins with change in step counts | 12 weeks
  Correlation of baseline proteins with change in step counts

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Hegde, MD, Principal Investigator — Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ngo D, Sinha S, Shen D, Kuhn EW, Keyes MJ, Shi X, Benson MD, O'Sullivan JF, Keshishian H, Farrell LA, Fifer MA, Vasan RS, Sabatine MS, Larson MG, Carr SA, Wang TJ, Gerszten RE. Aptamer-Based Proteomic Profiling Reveals Novel Candidate Biomarkers and Pathways in Cardiovascular Disease. Circulation. 2016 Jul 26;134(4):270-85. doi: 10.1161/CIRCULATIONAHA.116.021803. PMID 27444932
- [Background] Jacob J, Ngo D, Finkel N, Pitts R, Gleim S, Benson MD, Keyes MJ, Farrell LA, Morgan T, Jennings LL, Gerszten RE. Application of Large-Scale Aptamer-Based Proteomic Profiling to Planned Myocardial Infarctions. Circulation. 2018 Mar 20;137(12):1270-1277. doi: 10.1161/CIRCULATIONAHA.117.029443. Epub 2017 Dec 8. PMID 29222138
- [Background] Wallentin L, Eriksson N, Olszowka M, Grammer TB, Hagstrom E, Held C, Kleber ME, Koenig W, Marz W, Stewart RAH, White HD, Aberg M, Siegbahn A. Plasma proteins associated with cardiovascular death in patients with chronic coronary heart disease: A retrospective study. PLoS Med. 2021 Jan 13;18(1):e1003513. doi: 10.1371/journal.pmed.1003513. eCollection 2021 Jan. PMID 33439866
- [Background] Sanders-van Wijk S, Tromp J, Beussink-Nelson L, Hage C, Svedlund S, Saraste A, Swat SA, Sanchez C, Njoroge J, Tan RS, Fermer ML, Gan LM, Lund LH, Lam CSP, Shah SJ. Proteomic Evaluation of the Comorbidity-Inflammation Paradigm in Heart Failure With Preserved Ejection Fraction: Results From the PROMIS-HFpEF Study. Circulation. 2020 Nov 24;142(21):2029-2044. doi: 10.1161/CIRCULATIONAHA.120.045810. Epub 2020 Oct 9. PMID 33034202
- [Background] Santos-Parker JR, Santos-Parker KS, McQueen MB, Martens CR, Seals DR. Habitual aerobic exercise and circulating proteomic patterns in healthy adults: relation to indicators of healthspan. J Appl Physiol (1985). 2018 Nov 1;125(5):1646-1659. doi: 10.1152/japplphysiol.00458.2018. Epub 2018 Sep 20. PMID 30236049
- [Background] Stattin K, Lind L, Elmstahl S, Wolk A, Lemming EW, Melhus H, Michaelsson K, Byberg L. Physical activity is associated with a large number of cardiovascular-specific proteins: Cross-sectional analyses in two independent cohorts. Eur J Prev Cardiol. 2019 Nov;26(17):1865-1873. doi: 10.1177/2047487319868033. Epub 2019 Aug 14. PMID 31409108
- [Background] Contrepois K, Wu S, Moneghetti KJ, Hornburg D, Ahadi S, Tsai MS, Metwally AA, Wei E, Lee-McMullen B, Quijada JV, Chen S, Christle JW, Ellenberger M, Balliu B, Taylor S, Durrant MG, Knowles DA, Choudhry H, Ashland M, Bahmani A, Enslen B, Amsallem M, Kobayashi Y, Avina M, Perelman D, Schussler-Fiorenza Rose SM, Zhou W, Ashley EA, Montgomery SB, Chaib H, Haddad F, Snyder MP. Molecular Choreography of Acute Exercise. Cell. 2020 May 28;181(5):1112-1130.e16. doi: 10.1016/j.cell.2020.04.043. PMID 32470399
- [Background] Robbins JM, Peterson B, Schranner D, Tahir UA, Rienmuller T, Deng S, Keyes MJ, Katz DH, Beltran PMJ, Barber JL, Baumgartner C, Carr SA, Ghosh S, Shen C, Jennings LL, Ross R, Sarzynski MA, Bouchard C, Gerszten RE. Human plasma proteomic profiles indicative of cardiorespiratory fitness. Nat Metab. 2021 Jun;3(6):786-797. doi: 10.1038/s42255-021-00400-z. Epub 2021 May 27. PMID 34045743
- [Background] Shah AM, Claggett B, Loehr LR, Chang PP, Matsushita K, Kitzman D, Konety S, Kucharska-Newton A, Sueta CA, Mosley TH, Wright JD, Coresh J, Heiss G, Folsom AR, Solomon SD. Heart Failure Stages Among Older Adults in the Community: The Atherosclerosis Risk in Communities Study. Circulation. 2017 Jan 17;135(3):224-240. doi: 10.1161/CIRCULATIONAHA.116.023361. Epub 2016 Nov 23. PMID 27881564
- [Background] Hieda M, Sarma S, Hearon CM Jr, Dias KA, Martinez J, Samels M, Everding B, Palmer D, Livingston S, Morris M, Howden E, Levine BD. Increased Myocardial Stiffness in Patients With High-Risk Left Ventricular Hypertrophy: The Hallmark of Stage-B Heart Failure With Preserved Ejection Fraction. Circulation. 2020 Jan 14;141(2):115-123. doi: 10.1161/CIRCULATIONAHA.119.040332. Epub 2019 Dec 23. PMID 31865771
- [Background] Hieda M, Sarma S, Hearon CM Jr, MacNamara JP, Dias KA, Samels M, Palmer D, Livingston S, Morris M, Levine BD. One-Year Committed Exercise Training Reverses Abnormal Left Ventricular Myocardial Stiffness in Patients With Stage B Heart Failure With Preserved Ejection Fraction. Circulation. 2021 Sep 21;144(12):934-946. doi: 10.1161/CIRCULATIONAHA.121.054117. Epub 2021 Sep 20. PMID 34543068
- [Background] O'Connor CM, Whellan DJ, Lee KL, Keteyian SJ, Cooper LS, Ellis SJ, Leifer ES, Kraus WE, Kitzman DW, Blumenthal JA, Rendall DS, Miller NH, Fleg JL, Schulman KA, McKelvie RS, Zannad F, Pina IL; HF-ACTION Investigators. Efficacy and safety of exercise training in patients with chronic heart failure: HF-ACTION randomized controlled trial. JAMA. 2009 Apr 8;301(14):1439-50. doi: 10.1001/jama.2009.454. PMID 19351941
- [Background] Whellan DJ, O'Connor CM, Lee KL, Keteyian SJ, Cooper LS, Ellis SJ, Leifer ES, Kraus WE, Kitzman DW, Blumenthal JA, Rendall DS, Houston-Miller N, Fleg JL, Schulman KA, Pina IL; HF-ACTION Trial Investigators. Heart failure and a controlled trial investigating outcomes of exercise training (HF-ACTION): design and rationale. Am Heart J. 2007 Feb;153(2):201-11. doi: 10.1016/j.ahj.2006.11.007. PMID 17239677
- [Background] Bozkurt B, Fonarow GC, Goldberg LR, Guglin M, Josephson RA, Forman DE, Lin G, Lindenfeld J, O'Connor C, Panjrath G, Pina IL, Shah T, Sinha SS, Wolfel E; ACC's Heart Failure and Transplant Section and Leadership Council. Cardiac Rehabilitation for Patients With Heart Failure: JACC Expert Panel. J Am Coll Cardiol. 2021 Mar 23;77(11):1454-1469. doi: 10.1016/j.jacc.2021.01.030. PMID 33736829
- [Background] Keteyian SJ, Ades PA, Beatty AL, Gavic-Ott A, Hines S, Lui K, Schopfer DW, Thomas RJ, Sperling LS. A Review of the Design and Implementation of a Hybrid Cardiac Rehabilitation Program: AN EXPANDING OPPORTUNITY FOR OPTIMIZING CARDIOVASCULAR CARE. J Cardiopulm Rehabil Prev. 2022 Jan 1;42(1):1-9. doi: 10.1097/HCR.0000000000000634. PMID 34433760
- [Background] Rawstorn JC, Ball K, Oldenburg B, Chow CK, McNaughton SA, Lamb KE, Gao L, Moodie M, Amerena J, Nadurata V, Neil C, Cameron S, Maddison R. Smartphone Cardiac Rehabilitation, Assisted Self-Management Versus Usual Care: Protocol for a Multicenter Randomized Controlled Trial to Compare Effects and Costs Among People With Coronary Heart Disease. JMIR Res Protoc. 2020 Jan 27;9(1):e15022. doi: 10.2196/15022. PMID 32012103
- [Background] Reeves GR, Whellan DJ, Duncan P, O'Connor CM, Pastva AM, Eggebeen JD, Hewston LA, Morgan TM, Reed SD, Rejeski WJ, Mentz RJ, Rosenberg PB, Kitzman DW; REHAB-HF Trial Investigators. Rehabilitation Therapy in Older Acute Heart Failure Patients (REHAB-HF) trial: Design and rationale. Am Heart J. 2017 Mar;185:130-139. doi: 10.1016/j.ahj.2016.12.012. Epub 2016 Dec 28. PMID 28267466